CLINICAL TRIAL: NCT02320032
Title: A Phase 1, Randomized, Open-Label Study Evaluating the Pharmacokinetics of Various Dosing Regimens of Aripiprazole Lauroxil in Subjects With Stable Schizophrenia
Brief Title: An Open-Label Study of Aripiprazole Lauroxil in Subjects With Stable Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK9072-A105
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
Keywords: Alkermes; Schizophrenia; Aripiprazole; Aripiprazole lauroxil; ALKS 9072
MeSH Terms: conditions — Schizophrenia | interventions — aripiprazole lauroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aripiprazole Lauroxil - A (Experimental): Intramuscular (IM) injection Dose and Dosing Sequence A
  Interventions: Drug: Aripiprazole Lauroxil
- Aripiprazole Lauroxil - B (Experimental): Intramuscular (IM) injection Dose and Dosing Sequence B
  Interventions: Drug: Aripiprazole Lauroxil
- Aripiprazole Lauroxil - C (Experimental): Intramuscular (IM) injection Dose and Dosing Sequence C
  Interventions: Drug: Aripiprazole Lauroxil
- Aripiprazole Lauroxil - D (Experimental): Intramuscular (IM) injection Dose and Dosing Sequence D
  Interventions: Drug: Aripiprazole Lauroxil

INTERVENTIONS:
Drug: Aripiprazole Lauroxil — Gluteal IM injection, given once every 4 to 8 weeks

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of various doses and dosing intervals of aripiprazole lauroxil.

ELIGIBILITY:
Inclusion Criteria:

* Has stable schizophrenia or schizoaffective disorder
* Has demonstrated ability to tolerate aripiprazole
* Has been on a stable antipsychotic medication regimen without any changes for at least 2 months prior to screening
* Has a body mass index (BMI) of 18.0 to 35.0 kg/m2, inclusive
* Additional criteria may apply

Exclusion Criteria:

* Is pregnant, breastfeeding, or is planning to become pregnant during the study period
* Has received aripiprazole lauroxil or IM depot aripiprazole within 6 months, or other long-acting, injectable antipsychotic medication within 3 months
* Is a danger to himself/herself at screening or upon admission
* Has a history of or positive test result for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Has a positive urine drug screen at screening or Day 1
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
AUC 0-last | Up to 45 weeks
  Area under the plasma-concentration time curve from time zero to the last quantifiable plasma concentration
C max | Up to 45 weeks
  Maximum plasma concentration
T max | Up to 45 weeks
  Time to maximum plasma concentration

SECONDARY OUTCOMES:
AUC 0-tau | Up to 45 weeks
  Area under the plasma-concentration time curve over the dose interval
Safety and tolerability will be measured by incidence of adverse events | Up to 45 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, MD, Study Director — Alkermes, Inc.
Locations (16):
- United States (16):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Oakland Park, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas

REFERENCES:
- [Result] Hard ML, Mills RJ, Sadler BM, Turncliff RZ, Citrome L. Aripiprazole Lauroxil: Pharmacokinetic Profile of This Long-Acting Injectable Antipsychotic in Persons With Schizophrenia. J Clin Psychopharmacol. 2017 Jun;37(3):289-295. doi: 10.1097/JCP.0000000000000691. PMID 28350572
- [Derived] Weiden PJ, Du Y, von Moltke L, Wehr A, Hard M, Marandi M, Walling DP. Pharmacokinetics, Safety, and Tolerability of a 2-Month Dose Interval Regimen of the Long-Acting Injectable Antipsychotic Aripiprazole Lauroxil: Results From a 44-Week Phase I Study. CNS Drugs. 2020 Sep;34(9):961-972. doi: 10.1007/s40263-020-00745-1. PMID 32621071
- [Derived] Hard ML, Mills RJ, Sadler BM, Wehr AY, Weiden PJ, von Moltke L. Pharmacokinetic Profile of a 2-Month Dose Regimen of Aripiprazole Lauroxil: A Phase I Study and a Population Pharmacokinetic Model. CNS Drugs. 2017 Jul;31(7):617-624. doi: 10.1007/s40263-017-0447-7. PMID 28597226